CLINICAL TRIAL: NCT07033780
Title: Optimization of Prefrontal Theta-Burst Stimulation to Treat Depression: A Bench to First-in-Human Study
Brief Title: Theta-Burst Stimulation to Treat Depression
Acronym: INSPiRE-D
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Brain Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024/116-01
Record Dates: First submitted 2025-01-06; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: TMS; TBS; iTBS; iTBS-sh; iTBS-c; iTBS-s; Sham iTBS; Spaced iTBS; Compressed iTBS; LTP; Long Term Potentiation; Theta-Burst Stimulation; Intermittent Theta Burst Stimulation; Transcranial Magnetic Stimulation; MDD; Major Depressive Disorder; Depression; Depressed individuals; Brain Plasticity; Dorsolateral Prefrontal Cortex; DLPFC; Motor Cortex; Neuroplasticity
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: This phase I clinical trial will employ a double-blind, randomized controlled cross-over design with two experimental iTBS conditions (iTBS-c and iTBS-s).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be completed under double-blind conditions: (1) Participants will be blind to the hypothesis and potential differences in outcomes between iTBS-c and iTBS-s; (2) The research staff conducting the clinical and TMS-EEG assessments will be blind to group assignment.
  Trained personnel administering iTBS (i.e., the interventionist) will not be blinded to the iTBS condition being administered. Therefore, trained personnel who administer iTBS will not be permitted to complete any study assessments following the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spaced iTBS (Experimental): Upon completion of Visits 1-2 (Screening and MRI), participants randomized to iTBS-s will complete a baseline TMS-EEG measurement, one iTBS-s intervention session, and post-iTBS TMS-EEG measurements in each of Visits 3-5. Following this, participants will undergo a washout period of at least two weeks. Then, participants will return to complete the opposite iTBS intervention across Visits 6-8. The procedures and visits will be identical, but the participant will receive the other iTBS intervention that they were not initially randomized to.
  Interventions: Device: Spaced iTBS
- Compressed iTBS (Active Comparator): Upon completion of Visits 1-2 (Screening and MRI), participants randomized to iTBS-c will complete a baseline TMS-EEG measurement, one iTBS-c intervention session, and post-iTBS TMS-EEG measurements in each of Visits 3-5. Following this, participants will undergo a washout period of at least two weeks. Then, participants will return to complete the opposite iTBS intervention across Visits 6-8. The procedures and visits will be identical, but the participant will receive the other iTBS intervention that they were not initially randomized to.
  Interventions: Device: Compressed iTBS

INTERVENTIONS:
Device: Spaced iTBS — Intermittent Theta-Burst Stimulation (iTBS) is a form of non-invasive brain stimulation that uses magnetic pulses applied to the scalp using a coil. iTBS will be used to stimulate the left dorsolateral prefrontal cortex (DLPFC) to enhance long-term potentiation (LTP)-like activity, a physiological mechanism associated with brain plasticity. TMS-EEG will be performed to measure changes in brain plasticity throughout the trial. An EEG cap will be placed on the participant's head, and the electrodes on the cap will be filled with saline gel using a dull syringe.
  During the intervention, the study team will conduct a baseline TMS-EEG measurement consisting of single TMS pulses. Participants will then complete iTBS-s (experimental study intervention), which will be delivered to the left DLPFC. Following iTBS-s, post-iTBS TMS-EEG measurements will be obtained consisting of 3 TMS trains delivered to the left DLPFC (Post-0, Post-20, and Post-60 minutes).
  Other Names: iTBS-s
  Arms: Spaced iTBS
Device: Compressed iTBS — Intermittent Theta-Burst Stimulation (iTBS) is a form of non-invasive brain stimulation that uses magnetic pulses applied to the scalp using a coil. iTBS will be used to stimulate the left dorsolateral prefrontal cortex (DLPFC) to enhance long-term potentiation (LTP)-like activity, a physiological mechanism associated with brain plasticity. TMS-EEG will be performed to measure changes in brain plasticity throughout the trial. An EEG cap will be placed on the participant's head, and the electrodes on the cap will be filled with saline gel using a dull syringe.
  During the intervention, the study team will conduct a baseline TMS-EEG measurement consisting of single TMS pulses. Participants will then complete iTBS-c (active comparator), which will be delivered to the left DLPFC. Following iTBS-c, post-iTBS TMS-EEG measurements will be obtained consisting of 3 TMS trains delivered to the left DLPFC (Post-0, Post-20, and Post-60 minutes).
  Other Names: iTBS-c
  Arms: Compressed iTBS

SUMMARY:
The goal of this clinical trial is to explore the effects of non-invasive brain stimulation protocols using intermittent theta-burst stimulation (iTBS) on brain plasticity and depression severity in depressed individuals aged 18 to 50 years old. Brain plasticity is the brain's ability to change through growth or reorganization. iTBS is a form of transcranial magnetic stimulation (TMS), where magnetic pulses are applied to the scalp using a coil. These pulses pass through the scalp, and can alter brain activity in the area underneath the coil. Based on previous research conducted in animals and humans, researchers believe that iTBS can strengthen the connections between cells in the brain, leading to improved brain plasticity.

This trial will compare the effects of the compressed iTBS (iTBS-c) protocol, which is commonly used to treat depression, and the spaced iTBS (iTBS-s) protocol. Researchers want to find out which protocol is better able to produce changes in brain plasticity and improve symptoms of depression among individuals diagnosed with Major Depressive Disorder (MDD). In this trial, participants will be randomized to receive 3 sessions of iTBS-s or iTBS-c, undergo a washout period of at least 2 weeks, then complete 3 sessions of the opposite iTBS intervention.

Participants will complete 5 study visits within the span of 2-3 months, including:

* Screening assessments to determine eligibility & 1 sham iTBS (iTBS-sh) session to assess tolerability of the brain stimulation (Visit 1);
* 1 Magnetic Resonance Imaging (MRI) brain scan and randomization (Visit 2);
* Safety and clinical assessments, iTBS-s or iTBS-c intervention, TMS evoked electroencephalography (TMS-EEG) measurements, and post-iTBS questionnaires (Visits 3-5) followed by a washout period of at least 2 weeks;
* Safety and clinical assessments, the opposite iTBS-s or iTBS-c intervention originally randomized to, TMS-EEG measurements, and post-iTBS questionnaires (Visits 6-8).

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a mental illness affecting millions of individuals worldwide and in Canada, and is a leading cause of morbidity, mortality, and disability. While antidepressant medications are effective in treating MDD, their efficacy is moderate and systemic side-effects persist, such as sexual dysfunction, drowsiness, weight gain, and dry mouth. Thus, more effective treatments are needed for MDD.

Neuroimaging techniques have implicated the dysregulation of brain plasticity in depression. In particular, long-term potentiation (LTP)-like activity in the dorsolateral prefrontal cortex (DLPFC) and the motor cortex is known to be impaired in MDD. As such, transcranial magnetic stimulation (TMS)-based interventions, which aim to modify underlying cortical activity, are now established treatments of depression. Intermittent theta-burst stimulation (iTBS), a novel form of repetitive TMS (rTMS) approved by the US Food and Drug Administration (FDA) for the treatment of depression, delivers intermittent, high-frequency theta bursts. It has been demonstrated to induce sustained plasticity in the DLPFC and the motor cortex. Studies have shown that iTBS is equally effective as conventional rTMS in terms of response rates, and its adverse effects are comparable to iTBS-sh and active rTMS. One key advantage of iTBS over rTMS is its time efficiency, with each session lasting approximately 3 min compared to up to 40 min with rTMS. Notwithstanding its efficiency, systematic reviews of RCTs indicate no significant difference in remission rates - defined as a reduction in symptoms below a threshold indicating euthymic state - between iTBS (~26%) and iTBS-sh (~19%), or between iTBS (32%) and rTMS (27%). Thus, while iTBS is well tolerated, efficient and effective in reducing symptoms of MDD, its efficacy is still far from optimal as is the case for other treatments of depression.

Based on promising research conducted in the hippocampus of rodents, the investigators believe that modifying some parameters of the iTBS protocol may be more effective in inducing plasticity than the currently used iTBS protocol. Thus, in this trial researchers aim to determine whether an optimized iTBS protocol will result in better LTP-like activity in the DLPFC of adults with MDD.

The objectives and hypotheses of the study are as follows:

Objective 1: To compare the ability of iTBS-c vs. iTBS-s to induce DLPFC LTP-like activity in depressed adults as measured using TMS-electroencephalography (EEG).

Hypothesis 1a: iTBS-s will induce stronger DLPFC LTP-like activity compared to iTBS-c.

Hypothesis 1b: iTBS-s will induce longer-lasting DLPFC LTP-like activity compared to iTBS-c.

Objective 2: To evaluate the relationship between DLPFC LTP-like activity and changes in depression severity, as measured by the Montgomery-Asberg Depression Rating Scale (MADRS).

Hypothesis 2a: DLPFC LTP-like activity will be inversely associated with baseline depressive symptoms.

Hypothesis 2b: DLPFC LTP-like activity will be associated with improvement in depressive symptoms on Visits 3 to 5.

Objective 3: To compare the effect of iTBS-c vs. iTBS-c within-subjects on DLPFC LTP-like activity in depressed adults as measured using TMS-EEG during the cross-over phase of the study.

Hypothesis 3: iTBS-s will induce stronger DLPFC LTP-like activity compared to iTBS-c within-subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50 years old;
* Must meet criteria for a current Major Depressive Episode (MDE) as ascertained using the Structured Clinical Interview for DSM 5 (SCID-5);
* Hamilton Rating Scale for Depression (HRSD-17) score > 7;
* Must be on a stable antidepressant regimen for a minimum of 4 weeks prior to enrollment, if currently taking antidepressants;
* Right handed or ambidextrous, assessed using the Edinburgh Handedness Inventory (EHI);
* Sufficiently proficient in English to complete the required study assessments, as per investigator judgement;
* Willingness and capacity to provide informed consent;
* Willingness to comply with all study procedures.

Exclusion Criteria:

* Age 17 years or less, or greater than 51 years old, as brain plasticity is known to be affected by age;
* Presence of any DSM-5 diagnosis (other than MDD), known to be associated with prefrontal cortical dysfunction, including lifetime diagnoses of bipolar disorder, intellectual disability, or a psychotic disorder, assessed using the SCID-5 and as per investigator judgement;
* Presence of acute suicidal intent, as determined by the Scale for Suicidal Ideation (SSI);
* Contradictions to MRI or TMS (e.g., cardiac pacemaker, acoustic device, history of seizures, pregnancy), assessed using the MRI Safety Form and TMS Adult Safety Screen (TASS) and as per investigator judgement;
* Left handed, assessed using the EHI, to minimize the heterogeneity in cortical excitability and plasticity;
* Current antipsychotic, antiepileptic, or benzodiazepine use given their potential effects on cortical plasticity, as ascertained through a medication review. An exception will be made if they are taking gabapentin or pregabalin prescribed only for chronic pain, and if the dose had been stable for at least 4 weeks prior to study enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
DLPFC LTP-like Activity - CEA Ratio at Visit 3 | Immediately before iTBS and at 20 and 60 minutes post-iTBS at Visit 3
  Cortical evoked activity (CEA) over the left DLPFC will be measured using TMS-EEG before the application of the iTBS condition and at 0, 20 and 60-minutes post-iTBS in Visit 3. The CEA ratio will be calculated by dividing the average post-iTBS CEA (across post-20 and post-60 minutes) by the pre-iTBS CEA. Hypothesis 1a will then be tested by comparing the CEA Ratio at Visit 3 between the group randomized to iTBS-s and the group randomized to iTBS-c.
DLPFC LTP-like Activity - Change in pre-iTBS CEA from Visit 3 to 4 | Pre-iTBS at Baseline (Visit 3) and Pre-iTBS at 24 hours post-baseline (Visit 4)
  Cortical evoked activity (CEA) over the left DLPFC will be measured using TMS-EEG before the application of the iTBS condition at Visit 3 (baseline), and again before iTBS at Visit 4 (24 hours post-baseline). Hypothesis 1b will be tested by comparing the change in pre-iTBS CEA from Visit 3 to Visit 4 between the group randomized to iTBS-s and the group randomized to iTBS-c.
DLPFC LTP-like Activity - Change in pre-iTBS CEA from Visit 4 to 5 | Pre-iTBS at 24 hours post-baseline (Visit 4) and Pre-iTBS at 6 days post-baseline (Visit 5)
  Cortical evoked activity (CEA) over the left DLPFC will be measured using TMS-EEG before the application of the iTBS condition at Visit 4 (24 hours post-baseline) and again before iTBS at Visit 5 (6 days post-baseline). Hypothesis 1b will be tested by comparing the change in pre-iTBS CEA from Visit 4 to Visit 5 between the group randomized to iTBS-s and the group randomized to iTBS-c.

SECONDARY OUTCOMES:
MADRS Scores - Hypothesis 2a | Visit 3 (baseline), Visit 4 (24 hours post-baseline), and Visit 5 (6 days post-baseline)
  Hypothesis 2a will be tested by comparing the association between the average CEA Ratio across Visits 3, 4, and 5 and baseline scores on the Montgomery-Åsberg Depression Rating Scale (MADRS), which ranges from 0 (minimum) to 60 (maximum), with higher scores reflecting greater depression severity.
MADRS Scores - Hypothesis 2b | Visit 3 (baseline), Visit 4 (24 hours post-baseline), and Visit 5 (6 days post-baseline)
  Hypothesis 2b will be tested by comparing the association between the CEA Ratio at each of Visits 3, 4, and 5 and the corresponding change in MADRS scores from baseline to post-iTBS at each visit.

OTHER OUTCOMES:
DLPFC LTP-like activity (within subjects) | After Visits 3-5 (first iTBS condition) and Visits 6-8 (second iTBS condition)
  To address Objective 3, the CEA Ratio will be calculated for each of Visits 3 through 8. The CEA ratios from Visits 3, 4, and 5 will be averaged to obtain the mean CEA Ratio for the first iTBS condition (iTBS-s or iTBS-c). Then, the CEA ratios from Visits 6, 7, and 8 will be averaged to determine the mean CEA Ratio for the other iTBS condition. The average CEA ratio of iTBS-s will be compared to the average CEA ratio of iTBS-c within subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pathophysiology of depression: the concept of synaptic plasticity — https://pubmed.ncbi.nlm.nih.gov/15177086/
- See also: Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial — https://pubmed.ncbi.nlm.nih.gov/20439832/
- See also: The role of neural plasticity in depression: from hippocampus to prefrontal cortex. Neural plasticity — https://pubmed.ncbi.nlm.nih.gov/28246558/
- See also: Impaired modulation of corticospinal excitability in drug-free patients with major depressive disorder: a theta-burst stimulation study — https://www.frontiersin.org/journals/human-neuroscience/articles/10.3389/fnhum.2019.00072/full
- See also: Efficacy of theta burst stimulation (TBS) for major depression: an exploratory meta-analysis of randomized and sham-controlled trials — https://pubmed.ncbi.nlm.nih.gov/28254709/
- See also: Theta-burst stimulation: A new form of TMS treatment for depression? Depression and anxiety — https://pubmed.ncbi.nlm.nih.gov/25450537/
- See also: Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression — https://pubmed.ncbi.nlm.nih.gov/8547583/
- See also: Theta burst stimulation for the acute treatment of major depressive disorder: a systematic review and meta-analysis — https://pubmed.ncbi.nlm.nih.gov/34050123/
- See also: Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial — https://pubmed.ncbi.nlm.nih.gov/29726344/